CLINICAL TRIAL: NCT01572584
Title: Accuracy of Lung Ultrasound in the Prediction of Pneumothorax Volume Assessed by CT Scan
Brief Title: Lung Ultrasound in the Evaluation of Pneumothorax Size
Acronym: LUS-PNXsize
Status: Completed | Type: Observational
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Giovanni Volpicelli, Medical Doctor, Department of Emergency Medicine, San Luigi Gonzaga Hospital
Other Study IDs: SLG-181/2011
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Pneumothorax
Keywords: Pneumothorax; Lung ultrasound; Chest sonography
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background

* Assessment of the percentage of lung collapse is crucial in the therapeutic decision-making of pneumothorax.
* The methods normally used to this purpose are radiological. Computerized tomography scan (CT) is highly accurate because it allows the exact evaluation of the volume of the air layer. However, in clinical practice assessment of the volume of pneumothorax mainly relies on the measurement of the inter-pleural distance at conventional chest radiography (CXR). This latter method is inaccurate.
* Lung ultrasound is a new method highly accurate in the first diagnosis of pneumothorax, with a sensitivity superior to CXR and similar to CT in case of traumatic pneumothorax.
* The scientific community is actually debating about the usefulness of lung ultrasound in the quantification of pneumothorax []. Lung ultrasound can assess the superficial extension of the pneumothorax, but cannot evaluate its volume.

Aim

* Main purpose of the study is to compare measurement of the superficial extension of pneumothorax on the chest wall obtained by lung ultrasound, to the evaluation of the air volume performed by CT in patients with pneumothorax.
* The main hypothesis of the study is that the cut-off between small (<11% of lung collapse) and large (>11% of lung collapse) pneumothorax can be identified by a lung ultrasound evaluation of the superficial extension of pneumothorax.
* Second purpose of the study is to compare the accuracies of lung ultrasound and CXR in predicting the volume of pneumothorax assessed by CT.
* Secondary hypothesis is that lung ultrasound demonstrates greater accuracy in the prediction of volume of pneumothorax and percentage of lung collapse.

Methods

* Patients with a diagnosis of pneumothorax confirmed at CT are prospectively enrolled and submitted to lung ultrasound within 20 min from the CT study.
* Different locations of the sonographic "lung point" on the chest wall (i.e. the point on the chest wall where the sonographic pattern of the normally aerated lung alternates with the pathologic sonographic pattern of pneumothorax) are compared with different volumes of pneumothorax measured by CT.

ELIGIBILITY:
Inclusion Criteria:

* Radiologic diagnosis of pneumothorax
* Clinical need to perform a CT scan
* Ability to perform the lung ultrasound imaging within 20 minutes from the CT study

Exclusion Criteria:

* age less than 16 years

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the Emergency Department Patients admitted to the Hospital Outpatients from the Radiology Department who undergo invasive thoracic procedures
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The ultrasound lung point on the thorax wall versus the volume of pneumothorax at CT scan | The ultrasound lung point that the best discriminates a pneumothorax volume more than 11%

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Volpicelli, MD, Principal Investigator — San Luigi Gonzaga Hospital
Locations (1):
- San Luigi Gonzaga University Hospital, Orbassano, Torino, Italy

REFERENCES:
- [Background] Blaivas M, Lyon M, Duggal S. A prospective comparison of supine chest radiography and bedside ultrasound for the diagnosis of traumatic pneumothorax. Acad Emerg Med. 2005 Sep;12(9):844-9. doi: 10.1197/j.aem.2005.05.005. PMID 16141018
- [Background] Soldati G, Testa A, Sher S, Pignataro G, La Sala M, Silveri NG. Occult traumatic pneumothorax: diagnostic accuracy of lung ultrasonography in the emergency department. Chest. 2008 Jan;133(1):204-11. doi: 10.1378/chest.07-1595. Epub 2007 Oct 9. PMID 17925411
- [Background] Reissig A, Kroegel C. Accuracy of transthoracic sonography in excluding post-interventional pneumothorax and hydropneumothorax. Comparison to chest radiography. Eur J Radiol. 2005 Mar;53(3):463-70. doi: 10.1016/j.ejrad.2004.04.014. PMID 15741021
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A. The "lung point": an ultrasound sign specific to pneumothorax. Intensive Care Med. 2000 Oct;26(10):1434-40. doi: 10.1007/s001340000627. PMID 11126253
- [Background] Baumann MH, Strange C, Heffner JE, Light R, Kirby TJ, Klein J, Luketich JD, Panacek EA, Sahn SA; AACP Pneumothorax Consensus Group. Management of spontaneous pneumothorax: an American College of Chest Physicians Delphi consensus statement. Chest. 2001 Feb;119(2):590-602. doi: 10.1378/chest.119.2.590. PMID 11171742
- [Background] Engdahl O, Toft T, Boe J. Chest radiograph--a poor method for determining the size of a pneumothorax. Chest. 1993 Jan;103(1):26-9. doi: 10.1378/chest.103.1.26. PMID 8417891
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031